CLINICAL TRIAL: NCT04487587
Title: A Randomised Double Blind Placebo Controlled Phase II Clinical Trial of Cediranib and Olaparib Maintenance in Advanced Recurrent Cervical Cancer (COMICE)
Brief Title: A Phase II Clinical Trial of Cediranib and Olaparib Maintenance in Advanced Recurrent Cervical Cancer
Acronym: COMICE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Clatterbridge Cancer Centre NHS Foundation Trust (Other)
Collaborators: University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCC844
Record Dates: First submitted 2020-02-12; First posted 2020-07-27 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — cediranib; olaparib

STUDY DESIGN:
Intervention Model Description: Patients are randomised 1:1 to either placebo Cediranib and Olaparib or active Cediranib and Olaparib
Who Masked: Participant, Care Provider, Investigator
Masking Description: COMICE is a double blind trial, the Investigator, Patient, Hospital Staff, Pharmacy and the COMICE trial team (Chief Investigator, Monitor, Trial Coordinator) are blinded to the treatment allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Cediranib 20mg tablet OD (5 days out of 7) and Olaparib 300mg tablet BD (continuous) + standard of care
  Interventions: Drug: Cediranib, Olaparib
- Placebo (Placebo Comparator): Placebo Cediranib 20mg tablet OD (5 days out of 7) and Placebo Olaparib 300mg tablet BD (continuous) + standard of care
  Interventions: Drug: Cediranib, Olaparib

INTERVENTIONS:
Drug: Cediranib, Olaparib — Cediranib film coated tablet, Olaparib film coated tablet

SUMMARY:
COMICE is a randomised, double blind placebo controlled Phase II trial. The trial is recruiting 108 patients with advanced recurrent cervical cancer who have completed their 1st line chemotherapy for advanced/recurrent disease. Patients will be randomised to either placebo Cediranib and Olaparib or active Cediranib and Olaparib and will remain on treatment until progression of disease, unacceptable toxicity or withdrawal of consent. Patients will be assessed for disease progression every 8 weeks through CT/MRI imaging. The primary end point is Progression Free Survival.

DETAILED DESCRIPTION:
Cervical cancer is the 4th most prevalent female cancer worldwide. In the UK there are around 3,207 new cases each year (2013) and 890 deaths (2012) (http://www.cancerresearchuk.org/health-professional/cancer-statistics/statistics-by-cancer-type/cervical-cancer). It is the most common cancer in females under 35 with the majority of cases diagnosed in women aged 25-64. There is a large unmet need for active treatments in metastatic and recurrent cervical cancer patients. Although early-stage and locally advanced cancers may be cured with radical surgery, chemoradiotherapy or both, there are limited options for patients with metastatic disease or persistent/ recurrent disease after platinum-based chemoradiotherapy. Patients treated with chemotherapy for metastatic or relapsed cervical cancer respond poorly to conventional chemotherapy (overall response rate [ORR] of 30-35%) with a median overall survival of less than a year. The recent publication of a phase III randomised controlled trial GOG 240 demonstrating a 3.7 month improvement in median overall survival with the addition of bevacizumab to combination chemotherapy has offered some hope for these patients. The ORR and progression free survival (PFS) were also improved in patients receiving bevacizumab compared to those receiving chemotherapy alone. The advantage seen with bevacizumab persisted in some subsets of patients including those aged 48-56 years, and those with recurrent /persistent disease. Bevacizumab was also effective in patients who had undergone pelvic irradiation. This was the first time a targeted agent had significantly improved OS in gynaecological cancer.

High tumour angiogenesis is associated with poor survival when cervical cancer is treated with radiotherapy and high tumour vascularity is a significant prognostic factor independent of tumour radiosensitivity. A relationship between vascular endothelial growth factor (VEGF) expression and OS has been demonstrated in patients treated with radiotherapy, and a review of multiple biomarker studies in cervix cancer has highlighted the importance of VEGF as an adverse prognostic factor. Targeting VEGF in cervical cancer may potentially exploit the role of human papilloma virus (HPV, particularly subtypes 16 and 18) in the causation of cervical cancer. The role of HPV in oncogenesis relates to the E6 and E7 proteins, with the former promoting degradation of p53 while E7 inactivates retinoblastoma protein. Degradation of p53 may be responsible for activation of angiogenesis through production of VEGF and downregulation of a potent angiogenesis inhibitor, thrombospondin.

Cediranib is a highly potent inhibitor of the tyrosine kinase activity of VEGF receptors 1-3 (VEGFR 1-3.) The recently published CIRCCa study demonstrated an increased PFS, VEGF-R receptor inhibition and response rate with the addition of cediranib to carboplatin and paclitaxel chemotherapy. This was accompanied by a manageable increased toxicity (specifically diarrhoea and hypertension) with no detriment to QOL. The median PFS was 35weeks and 29 weeks in the cediranib and placebo arms respectively (HR 0.58 p= 0.032). Understanding which patients are most likely to derive benefit from these agents requires further evaluation as a priority.

Poly (ADP-ribose) polymerase (PARP) inhibitors including Olaparib may have potential activity in cancers deficient in DNA repair genes or signalling pathways that mitigate DNA repair. PARP inhibitors have demonstrated selectivity for cells harbouring homologous recombination (HR) deficiencies such as those with BRCA mutations. HR deficient cells are unable to maintain genomic integrity in the presence of large numbers of DNA DSBs and are therefore sensitive to PARP inhibition. The activity of PARP inhibitors in not limited to those with BRCA mutations and may demonstrate synthetic lethality in cancers deficient in other proteins mitigating DNA repair, such as those with mutations in Fanconi anaemia complementation group (FANC) proteins. Thus synthetic lethality may be more broadly applied to cancers with an impaired HR pathway.

It is well recognised that persistent genital infection with high risk strain(s) of HPV is necessary for the development of cervical cancer. Cells expressing high risk HPV oncoproteins (E6 and E7, see above) demonstrate increased levels of DNA damage and chromosomal instability, which may be a consequence of replicative stress; a process which is associated with a number of cancer-prone syndromes. There is also evidence that HPV oncoproteins inhibit the activation of DNA repair checkpoints, promote inappropriate DNA repair checkpoint recovery and inhibit the activation of DNA repair mechanisms.

Current therapeutic modalities for cervical cancer exploit the sensitivity of these tumours to DNA damaging agents such as ionising radiation and platinum chemotherapeutic agents. Poly (ADP-ribose) polymerase (PARP) inhibitors reduce the DNA repair capacity of cells and can induce synthetic lethality in cancers with underlying defects in DNA repair mechanisms such as BRCA mutations (Scott, Swisher, and Kaufmann 2015). The investigators therefore postulate that the action of HPV oncoproteins will lead to increase rates of DNA damage and reduced efficiency of DNA repair, leading in turn to increased susceptibility to PARP inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Histologically proven carcinoma of the cervix (squamous, adenocarcinoma or mixed adeno/squamous).
* Completion of first line platinum-based chemotherapy for advanced /recurrent disease, leading to either a complete response, partial response or stable disease.
* ECOG performance status 0 or 1
* Randomisation within 8 weeks of completion of chemotherapy
* Patients may have received previous chemoradiotherapy and neoadjuvant chemotherapy given with a curative intent.
* Creatinine Clearance ≥ 51mls/min
* Adequate haematological and biochemical function, as follows:
* Haemoglobin > 10g/dl (with no blood transfusion in the 28 days prior to randomisation) Neutrophils > 1.5 x 109/l
* Platelets > 100 x 109/l
* Bilirubin < 1.5 x ULN
* ALT or AST/ SGOT < 3 x ULN (or ≤5 x ULN if hepatic metastases present)
* Alkaline Phosphatase < 3 x ULN (or ≤5 x ULN if hepatic metastases present)
* Adequate coagulation, as follows:
* Prothrombin ratio (PTR) / INR ≤ 1.5 or
* PTR / INR between 2.0 and 3.0 for patients on stable doses of anticoagulants
* Partial thromboplastin time <1.2 x control
* Life expectancy >12 weeks.
* Informed written consent
* Contrast enhanced computerised tomography (CT) scan or magnetic resonance imaging (MRI) of the abdomen and pelvis and a CT scan of the chest within 28 days prior to commencing randomisation (with RECIST 1.1)
* Adequately controlled thyroid function, with no symptoms of thyroid dysfunction
* Able to swallow and retain oral medications and without gastrointestinal (GI) illnesses that would preclude absorption of cediranib or olaparib

Exclusion Criteria:

* Disease that is potentially treatable with exenterative surgery.
* Relapse confined to the pelvis after radical surgery in circumstance where radiotherapy or chemoradiotherapy would be appropriate.
* More than one line of prior chemotherapy for advanced/recurrent disease. Neoadjuvant chemotherapy is not counted.
* Prior treatment with anti-angiogenic agents (with the exception of bevacizumab given as part of first line chemotherapy)
* Persisting ≥Grade 2 CTCAE from previous anti-cancer previous systemic anti-cancer therapy except haematological toxicity (see inclusion criteria "Adequate haematological function") and alopecia.
* History of other malignancy within the previous 5 years except for:
* Curatively treated basal cell or squamous cell carcinoma of skin; in situ cancer of the cervix, ductal carcinoma in situ of the breast or stage 1, grade 1 endometrial carcinoma.
* Curatively treated other solid tumors including lymphomas (without bone marrow involvement) with no evidence of disease for ≥5 years prior to start of IMPs.
* Pregnant or lactating women.
* Fertile woman of childbearing potential not willing to use adequate contraception (oral contraceptives, intrauterine device or barrier method of contraception in conjunction with spermicidal jelly or surgically sterile) for the study duration and at least six months afterwards
* Evidence of uncontrolled infection. (Defined as infection that cannot be resolved readily with antibiotics prior to patient entry into the trial for example a pelvic collection)
* History of pelvic fistulae.
* History of abdominal fistula that has been surgically corrected within 6 months of starting treatment. Patient should be deemed low risk of recurrent fistula
* Sub-acute or acute intestinal obstruction.
* Major surgery within 28 days or anticipated while on study.
* Non-healing wound, ulcer or bone fracture.
* Active bleeding.
* History or evidence of thrombotic or haemorrhagic disorders.
* History of stroke or transient ischemic attack within 6 months
* Proteinuria > 1+ on dipstick on two consecutive dipsticks taken no less than 1 week apart, unless urinary protein is <1.5g in a 24 hour period.
* Significant cardiovascular disease (arterial thrombotic event within 12 months, uncontrolled hypertension, myocardial infarction or angina within 6 months, NYHA grade 2 or worse congestive cardiac failure, grade ≥ 3 peripheral vascular disease or cardiac arrhythmia requiring medication). Patients with rate-controlled atrial fibrillation are eligible.
* Prolonged QTc (corrected) interval of >470ms on ECG or a family history of long QT syndrome.
* Patients with symptomatic uncontrolled brain or meningeal metastases CNS disease (brain metastases, uncontrolled seizures or cerebrovascular accident/transient ischaemic attack /subarachnoid haemorrhage within 6 months).
* (A scan to confirm the absence of brain metastases is not required)
* A history of poorly controlled hypertension or resting BP>140/90 mmHG in the presence or absence of a stable regimen of anti-hypertensive therapy (measurements will be made after the patient has been resting supine for a minimum of 5 minutes. Two or more readings should be taken at 2 minute intervals and averaged. If the first two diastolic readings differ by more than 5mmHG, then an additional reading should be obtained and averaged).
* History of significant gastrointestinal impairment. Defined as active inflammatory bowel disease, bowel obstruction or any condition judged by the investigator to adversely impact on drug absorption or within 3 months prior to starting treatment.
* Patients with myelodysplastic syndrome/acute myeloid leukaemia.
* Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contra-indicates the use of an investigational drug or puts the patient at high risk for treatment-related complications.
* Patients who have been treated with potent inhibitors of CYP3A4 and 2C8 such as amiodaraone, clarithromycin, erythromycin, simvastatin, atorvastatin, lovastatin, montelukast sodium, verapamil, ketoconazole, miconazole, indinovir (and other antivirals) and diltiazem within 2 weeks of the first planned dose of cediranib will be excluded [NB These drugs are also prohibited during trial period]
* Patients treated with CYP3A inhibitors itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). Within 2 weeks of the first planned dose for strong inhibitors, and at least 1 week for moderate inhibitors.
* Concomitant use of known strong CYP3A inducers (e.g., phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). The required washout period prior to starting study treatments is 5 weeks for enzalutamide or phenobarbital and 4 weeks for other agents. [NB These drugs are also prohibited during trial period]
* Left ventricular ejection fraction (LVEF) < lower limit of normal (LLN) per institutional guidelines, or <55%, if threshold for normal not otherwise specified by institutional guidelines, for patients with the following risk factors:
* prior anthracycline, trastuzumab , chest radiotherapy, history of myocardial infarction within 6 months prior to start of study drug or other significant impaired cardiac function within 6-12 months prior to start of IMPs
* Patients who are known to be serologically positive for Hepatitis B, Hepatitis C or HIV, or who are receiving immunosuppressive treatment (with the exception of stable doses of steroids equivalent or less than prednisolone 10mg daily).
* History of intra-abdominal abscess within 3 months prior to starting treatment.
* Uncontrolled intercurrent illness including, but not limited to known ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or psychiatric illness/social situations that would limit compliance with study requirements.
* Prior allogeneic bone marrow transplant or double umbilical cord blood transplantation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — patients are eligible if diagnosed with cervical cancer
Enrollment: 79 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | The study ends when the last patient recruited has completed a minimum of 7 months on study. Recruitment period is 14 months so the maximum time a patient will be on study for is 21 months
  Date of disease progression
  *Current standard of care in this group of patients would be clinical follow up with no treatment

SECONDARY OUTCOMES:
Rate of Toxicity | SAEs are reported from randomisation to 30 days following the last administration of study IMP
  Safety (Toxicity, Serious Adverse Events)
Quality of Life FACT-Cx | completed at baseline then at the four weekly treatment review visit, up to the earlier of disease progression or 7 months
  Functional Assessment of Cancer Therapy- Cervical Cancer questionnaire
Overall Survival | from randomisation until date of death from any cause, assessed up to 21 months
  Date of death
Tumour Response | from date of randomisation until the date of first documented disease progression, assessed up to 21 months
  Tumour Response using RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Clatterbridge Cancer Centre, Metropolitan Borough of Wirral, United Kingdom

IPD SHARING:
Plan to Share IPD: No